CLINICAL TRIAL: NCT04152148
Title: A Phase I Clinical Trial of BAT4306F (for Injection) on Safety, Tolerability and Pharmacokinetics for Patients With CD20-positive, B-cell Non-Hodgkin's Lymphoma
Brief Title: A Phase I Clinical Trial of BAT4306F on Safety, Tolerability and Pharmacokinetics for Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT4306F-001-CR
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 500mg BAT4306F (Experimental): 3 weeks of a cycle
  Interventions: Biological: 500mg BAT4306F
- 750mg BAT4306F (Experimental): 3 weeks of a cycle
  Interventions: Biological: 750mg BAT4306F
- 900mg BAT4306F (Experimental): 3 weeks of a cycle
  Interventions: Biological: 900mg BAT4306F
- 1000mg BAT4306F (Experimental): 3 weeks of a cycle
  Interventions: Biological: 1000mg BAT4306F

INTERVENTIONS:
Biological: 500mg BAT4306F — Phase 1 dose titration study from BAT4306F 500mg to 1000mg, then choose a proper dose for amplification study based on DLT result
  Arms: 500mg BAT4306F
Biological: 750mg BAT4306F — Phase 1 dose titration study from BAT4306F 500mg to 1000mg, then choose a proper dose for amplification study based on DLT result
  Arms: 750mg BAT4306F
Biological: 900mg BAT4306F — Phase 1 dose titration study from BAT4306F 500mg to 1000mg, then choose a proper dose for amplification study based on DLT result
  Arms: 900mg BAT4306F
Biological: 1000mg BAT4306F — Phase 1 dose titration study from BAT4306F 500mg to 1000mg, then choose a proper dose for amplification study based on DLT result
  Arms: 1000mg BAT4306F

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of BAT4306F in patients with CD20-positive B-cell lymphoma

DETAILED DESCRIPTION:
1. The primary objective of the study is to evaluate the safety and tolerability of BAT4306F in patients with CD20-positive B-cell lymphoma, when the injection dosage escalates, to ultimately determine the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and recommended dosage for phase II clinical studies ( RP2D);
2. To evaluate the pharmacokinetics (PK) of BAT4306F(for injection);
3. To evaluate the immunogenicity profile of BAT4306F(for injection);
4. To evaluate the efficacy profile of BAT4306F (for injection);Using the Lugano criteria (2014), the 2008 IWCLL efficacy evaluation criteria, and the 2014 IWWM-7 efficacy evaluation criteria were used to evaluate the efficacy of related diseases at week 7, week 13, and week 19. The index of evaluation was ORR (including CR, PR, SD and PD, ORR is the proportion of patients with CR and PR).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry subjects must satisfy all of the following criteria: 1. Must be willing to provide written consent 2. Male or female, 18 years old or older 3. Histopathology test confirmed CD20-positive patients with relapsed/refractory/progressive non-Hodgkin's lymphoma, who have been treated with at least one course of standard anti-tumor regimen; 4. Has at least one measurable lesion: CLL patient monoclonal B cells≥5x 10^9/L. IgM in WM patients is greater than 2 times of the upper limit of normal. In patients other than CLL and WM, any diameter of the lymph node lesion ≥1.5cm or any extranodal lesion >1cm; 5. If the previous radiotherapy and chemotherapy cause toxic side effects, it needs to be restored to at least level 1 or returned to the baseline value or to be judged as irreversible (except for neurotoxicity related to grade 2 alopecia or platinum-containing treatment); 6. The patient's ECOG score was 0-2 points; 7. Expected survival is at least 6 months; 8. Subjects must have appropriate organ function and meet all of the following laboratory findings prior to enrollment: 1) The bone marrow reserve was basically normal: neutrophils (ANC) ≥ 1.0 × 10^9/L, hemoglobin (HB) ≥ 70 g/L, platelets (PLT) ≥ 50×10^9/L (Except for bone marrow invasion, B-NHL-related autoimmune cytopenia. bone marrow invasion will be judged by bone marrow biopsy, bone marrow smear, and bone marrow flow cytology results.) 2) Liver function is basically normal: ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN, TBIL ≤ 1.5×ULN (except for liver invasion. Patients with B-NHL-related autoimmune hemolytic anemia, TBIL is not subject to this limit); 3) Renal function is basically normal: creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 60mL/min; 4) The conventional coagulation examinations is basically normal: INR ≤ 1.5×ULN, APTT does not exceed the normal reference for 10 seconds; 9. Fertile female must be tested negative for serum pregnancy test; 10. If the patient is a male, it must be a male who has undergone surgical birth control, or use of an effective contraceptive method during the study period and within 12 months after the study drug is discontinued. In the case of female, an effective contraceptive procedure must be taken or during menopause or use of an effective contraceptive method during the study period and within 12 months of the study drug discontinuation, and avoid breastfeeding during the study period and within 12 months of the study drug discontinuation.

Exclusion Criteria:

Subjects will be excluded from the study if one or more of the following criteria are applicable: 1. Treatment with any monoclonal antibody within 3 months prior to the first dose; 2. Have used any anti-cancer vaccine in the past, or have used the HPV vaccine within 3 months prior to the study; 3. Used anti-CD20 mAb within 3 months prior to the first dose; 4. Radioimmunotherapy was used within 3 months prior to the first dose; 5. Treatment of transfusion, erythropoietin, granulocyte colony-stimulating factor or granulocyte-macrophage colony-stimulating factor within 2 weeks prior to the first dose; 6. Hematopoietic stem cell transplantation was performed 3 months before the first administration or hematopoietic stem cell transplantation was planned in 3 months; 7. A history of severe allergic reactions to humanized or murine monoclonal antibodies. (or is high reactivity / allergy to murine-derived products); 8. Evidence or medical history of central nervous system invasion or cranial neuropathy; 9. Concurrent with other malignant tumors (except for in situ cervical cancer, skin cancer, complete remission > 5 years of breast cancer and melanoma); 10. Other serious, uncontrollable concomitant diseases, including but not limited to: active infections, uncontrolled diabetes, uncontrollable hypertension, etc.; 11. Major surgery performed within 4 weeks prior to the first dose or during the expected study period, or if the surgical wound is not healed; 12. Patients with rheumatoid arthritis, granulomatous vasculitis, microscopic polyangiitis, toxic epidermal necrolysis or Stevens-Johnson syndrome; 13. Patients with chronic idiopathic bowel disease (including history of Crohns disease and Ulcerative Colitis), with intestinal obstruction or with chronic diarrhea; 14. Other past history, acute or chronic disease, mental illness, or laboratory test abnormalities that may result in increased risk of involvement in study or study drug administration, or interference in interpretation of research findings; 15. Pregnant or lactating women; 16. Received treatment in another clinical study within 4 weeks prior to the first dose; 17. Patients receiving high-dose corticosteroids (prednisolone greater than 10 mg/day or equivalent dosage of other drugs for 2 weeks or more) within 4 weeks prior to the first dose; 18. Virological examination: HBsAg positive; HBcAb positive and HBV-DNA detection ≥ detection upper limit; HCV antibody positive; HIV antibody positive; syphilis infection positive. 19. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | 4 weeks
  Safety and tolerability endpoint
Maximum tolerated dosed (MTD) | 4weeks
  Safety and tolerability endpoint
pharmacokinetics (PK) | up to 154 Days
  evaluate the pharmacokinetics (PK) of Recombinant Glycosylation-modified Anti-human-CD20 Monoclonal Antibody Solution for injection
CD19+ B lymphocyte ratio | up to 154 Days
  Pharmacodynamics endpoint
anti drug antibodies (ADA) | up to 154 Days
  Plasma level of anti drug antibodies (ADA) and neutralizing anti-drug antibodies (NADA) correlated with bevacizumab plasma level
ORR | the 7th week,the 13th week,the 19th week
  Overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, investigator, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided